CLINICAL TRIAL: NCT05407532
Title: Effectiveness of Oral Management Strategies on Improving Oral Frailty and Oral Bacteria Among Middle-aged and Elderly Hospitalized Adults With Pneumonia
Brief Title: Effectiveness of Oral Management Strategies on Improving Oral Frailty and Oral Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chen, Yen-Chin, Vice Head Nurse and Clinical Assistant Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: A-ER-110-281
Record Dates: First submitted 2022-01-27; First posted 2022-06-07 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Oral Hygiene; Pneumonia, Bacterial
Keywords: Pneumonia; Oral frailty; Oral bacteria; Oral management
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia | interventions — Population Groups; Therapeutics

STUDY DESIGN:
Intervention Model Description: 90 patients will be recruited and randomly assigned to three groups: the oral care group, the oral management group, and the standard care group.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group with oral care (Experimental): The investigators taught and monitored patients or caregivers to do oral care after meals and before sleep.
  Interventions: Procedure: Group with oral care
- Group with oral management (Experimental): The investigators taught and monitored patients or caregivers to oral health care plus oral exercises such as salivary glands massage methods after meals and before sleep.
  Interventions: Procedure: Group with oral management
- Group with standard of care (No Intervention): Only provided oral care education.

INTERVENTIONS:
Procedure: Group with oral management — The investigators provided information on oral health care plus oral exercises before meals, including salivary glands massage methods.
  Arms: Group with oral management
Procedure: Group with oral care — The investigators taught and monitored patients or caregivers to do oral care after meals and before sleep.
  Arms: Group with oral care

SUMMARY:
The aim of this study is to examine the effectiveness of nurse-driven oral management for improvements of oral frailty, and oral bacteria pneumonia patients with oral frailty using a randomized controlled trial (RCT) design. Hospitalized pneumonia patients (N = 90) will be randomized into three groups (oral management, oral care, and standard of care). The primary outcomes include the oral frailty measures determined by seven-item included oral hygiene, oral dryness, occlusion force, tongue-lip motor function, tongue pressure, mastication function, and swallowing function. Saliva samples were collected from the oral cavity before the bacterial culture was performed in the laboratory. Oral frailty measures and the presence of bacterial exposure were evaluated at baseline (1st day), on days 5, and at the time of discharge. The investigators will perform statistical analyses according to the intention-to-treat principle. All missing values will be imputed using the last value carry-forward method. The between-group differences will be examined using a mixed model in which group and time interaction will be included. This study finding could provide oral management strategies that could improve oral frailty and decrease oral bacteria for preventing recurrent pneumonia infection among middle-aged and older adults with pneumonia.

DETAILED DESCRIPTION:
The inclusion criteria will be as follows: (1) patients should be ≥ 50 years old; (2) patients' oral frailty should have been diagnosed with pneumonia, and (3) patients should have a Glasgow coma index of 15 points and be able to cooperate. Alternatively, the exclusion criteria will be as follows: (1) people with healthcare-related pneumonia; (2) those with head and neck cancer; or (3) those having an abnormal oral structure.

ELIGIBILITY:
Inclusion Criteria:

* Older than 50 years of age and equal
* Having mental clarity (Glasgow coma scale: 15)

Exclusion Criteria:

* A brief hospitalization (≤ 3 days) for non-acute care, such as uncomplicated elective percutaneous coronary intervention;
* Acute psychiatric syndromes;
* Received dental treatment in the last 6 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
oral frailty measures | The first day of admission (baseline value)
  The investigators measured seven items for patients to identify oral frailty including 1) the number of teeth, 2) masticatory ability, 3) difficulty making the "ta" sound, 4) tongue pressure, 5) abnormal swallowing pressure, and 6) tongue coating index (TCI), 7) oral dryness. Oral frailty was determined into three groups: non-oral frailty, 0 points; pre-oral frailty, 1-2 points; and oral frailty, ≥ 3 points.
Clearance of pneumonia associated oral bacteria | The first day of admission (baseline value)
  The investigators collected participants' gargling water for bacterial isolation and identification. The investigators asked the participant to gargle with 20 ml of N/S for approximately 20 seconds. The standard procedure for gargling was full mouth at least three times. The investigators collected gargling water in a bacterial collection bottle and sent it for bacterial culture within 2 hours. Bacterial colonies were quantified (CFU/ml). To observe the variation due to the different rinse solutions, the number of bacteria was determined again after the intervention. The investigators assessed the clearance of bacteria based on the baseline.
oral frailty measures | Day 5 of admission
  The investigators measured seven items for patients to identify oral frailty including 1) the number of teeth, 2) masticatory ability, 3) difficulty making the "ta" sound, 4) tongue pressure, 5) abnormal swallowing pressure, and 6) tongue coating index (TCI), 7) oral dryness. Oral frailty was determined into three groups: non-oral frailty, 0 points; pre-oral frailty, 1-2 points; and oral frailty, ≥ 3 points.
oral frailty measures | Discharge day
  The investigators measured seven items for patients to identify oral frailty including 1) the number of teeth, 2) masticatory ability, 3) difficulty making the "ta" sound, 4) tongue pressure, 5) abnormal swallowing pressure, and 6) tongue coating index (TCI), 7) oral dryness. Oral frailty was determined into three groups: non-oral frailty, 0 points; pre-oral frailty, 1-2 points; and oral frailty, ≥ 3 points.
Clearance of pneumonia associated oral bacteria | Discharge day
  The investigators collected participants' gargling water for bacterial isolation and identification. The investigators asked the participant to gargle with 20 ml of N/S for approximately 20 seconds. The standard procedure for gargling was full mouth at least three times. The investigators collected gargling water in a bacterial collection bottle and sent it for bacterial culture within 2 hours. Bacterial colonies were quantified (CFU/ml). To observe the variation due to the different rinse solutions, the number of bacteria was determined again after the intervention. The investigators assessed the clearance of bacteria based on the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: I-Yin Ho, Study Chair — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan, Tainan, Taiwan (r.o.c), Taiwan

REFERENCES:
- [Background] Chiang TC, Huang MS, Lu PL, Huang ST, Lin YC. The effect of oral care intervention on pneumonia hospitalization, Staphylococcus aureus distribution, and salivary bacterial concentration in Taiwan nursing home residents: a pilot study. BMC Infect Dis. 2020 May 27;20(1):374. doi: 10.1186/s12879-020-05061-z. PMID 32460697
- [Background] Minakuchi S, Tsuga K, Ikebe K, Ueda T, Tamura F, Nagao K, Furuya J, Matsuo K, Yamamoto K, Kanazawa M, Watanabe Y, Hirano H, Kikutani T, Sakurai K. Oral hypofunction in the older population: Position paper of the Japanese Society of Gerodontology in 2016. Gerodontology. 2018 Dec;35(4):317-324. doi: 10.1111/ger.12347. Epub 2018 Jun 8. PMID 29882364